CLINICAL TRIAL: NCT02185183
Title: Phase 2 Clinical Trial for Oral Administration of Alequel for Patients With IBD
Brief Title: Oral Administration of AlequelTM for Patients With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: YI2014-HMO-CTIL
Record Dates: First submitted 2014-04-28; First posted 2014-07-09 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2008-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- AlequelTM (Experimental): AlequelTM
  Interventions: Drug: Alequel

INTERVENTIONS:
Drug: Alequel — Alequel

SUMMARY:
Oral administration of Alequel, a mixture of proteins derived from the patient's bowel will be tested in patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
Oral administration of Alequel prepared from patients biopsies will be tested in patients with inflammatory bowel disease to determine its anti inflammatory effect.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease

Exclusion Criteria:

* Immune suppression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, M.D., Study Director — Hadassah Medical Organization

RESULTS

PARTICIPANT FLOW:
Groups:
- AlequelTM 30 ng Once a Day Orally: AlequelTM 30 ng once a day orally
  Alequel: Alequel
Period: Overall Study
Arm/Group | AlequelTM 30 ng Once a Day Orally
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AlequelTM
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 35 [26 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants] — 14 participants followed for improvement of disease
  participants
    Israel | 14
Crohn's disease activity index [Mean (Full Range); unit: units on a scale] — On a sclae of 100 to 400, a decrease in the score suggests improvement of disease activity
  units on a scale | 303 [100 to 400]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved in Disease Activity
Time Frame: 15 weeks
Measure: Number; unit: participants
Arm/Group | AlequelTM
Number analyzed (Participants) | 14
participants | 0

ADVERSE EVENTS:
Arm/Group | AlequelTM
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No